CLINICAL TRIAL: NCT03953157
Title: Improving Health of Women on Aromatase Inhibitors
Brief Title: Dietary and Exercise Interventions in Reducing Side Effects in Patients With Stage I-IIIa Breast Cancer Receiving Aromatase Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-001926; NCI-2019-02909 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Arthralgia; Postmenopausal; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8
MeSH Terms: conditions — Arthralgia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (dietary intervention) (Experimental): Patients receive a controlled anti-inflammatory diet over 12 weeks.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Questionnaire Administration
- Arm II (exercise intervention) (Experimental): Patients undergo controlled exercise sessions with a dedicated trainer 3 times a week for up to 1 hour each over 12 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Receive dietary intervention
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (dietary intervention)
Behavioral: Exercise Intervention — Receive exercise intervention
  Arms: Arm II (exercise intervention)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I/II trial studies how well dietary and exercise interventions work in reducing side effects in patients with stage I-IIIa breast cancer taking aromatase inhibitors. Anti-inflammatory Mediterranean dietary and bone strengthening exercise interventions may alleviate medication side effects such as joint and bone pain and protectively influence bone mineral density, improve heart functioning, and reduce risk of breast cancer recurrence in breast cancer patients taking aromatase inhibitors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To recruit an ethnically, racially and culturally diverse sample of postmenopausal women diagnosed with estrogen receptor positive breast cancer who are currently taking aromatase inhibitor (AI), establish eligibility, and randomly allocate 20 participants to a two-arm parallel intervention trial.

II. Conduct baseline measurements of: body composition and bone mineral density, reported muscle and joint pain; inflammatory, cardiovascular and bone health markers contained in blood serum; and, cardiovascular function.

III. Conduct a three month anti-inflammatory dietary intervention in one arm, and bone strengthening exercise intervention in the other study arm.

IV. At completion of these 3-month interventions, evaluate changes since baseline of body composition, bone density, reported muscle and joint pain, and inflammatory and cardiovascular measurements within each intervention arm, and preliminarily contrast changes between intervention arms.

V. Utilize results from both intervention arms to design a larger 2x2 randomized factorial trial designed to assess effects of anti-inflammatory diet, effects of bone promoting exercise, and combined diet and exercise intervention effects on joint and muscle pain, inflammatory markers, bone mineral density, and cardiovascular measures.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive a controlled anti-inflammatory diet over 12 weeks.

ARM II: Patients undergo controlled exercise sessions with a dedicated trainer 3 times a week for up to 1 hour each over 12 weeks.

After completion of study, patients are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months since breast cancer diagnosis up to 2 years since diagnosis.
* Diagnosed with localized breast cancer, up to stage IIIa.
* Has been taking aromatase inhibitor (AIs) for at least six months.
* Has been experiencing mild to moderate arthralgia (joint pain) for at least 2 months determined by the Brief Pain Inventory (BPI).
* At least 6 months post chemotherapy or radiation treatment.
* Subjects must be in good health as determined by medical history, physical examination, iDXA scan and clinical laboratory measurements.
* Postmenopausal either natural or surgical or postmenopausal caused by ovarian suppression treatments administered to premenopausal women.
* Currently taking aromatase inhibitor medication.

Exclusion Criteria:

* Diagnosed with metastatic breast cancer.
* Currently undergoing chemotherapy or radiation treatment.
* Food allergies of any kind, or any medical condition requiring mandatory dietary restrictions.
* A bone mineral density (BMD) T score less than -1, or fracture since taking AIs, or current use of glucocorticoids.
* Taking bisphosphonates or any other medication for bone loss.
* Significant cardiac, pulmonary, renal, liver or psychiatric disease.
* Currently undergoing or engaging in a regular exercise program.
* Muscular, orthopedic, or cardiovascular limitations that would prevent full participation in exercise.
* Body mass index (BMI) greater than 40 kg/m^2.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | Baseline up to 1 week post intervention
  Will be scanned by dual x-ray absorptiometry (iDXA).
Joint and muscle pain | Baseline up to 1 week post intervention
  Joint and muscle pain will be measured by the Brief Pain Inventory, a frequently administered assessment for studies of women on aromatase inhibitors (AIs). Participants will be asked about use of pain medication and supplements such as chondroitin and glucosamine. Subjects will also fill out standard visual analog scales to rate intensity of pain ranging from 1 to 10, as well as locate source of pain on standardized human figures available from International Society of Anesthetic Pharmacology. Additionally grip strength, a common marker of functional muscle and joint weakness, will be assessed using a dynamometer.
Inflammatory markers | Baseline up to 1 week post intervention
  Fasting blood samples will be collected at baseline and end of intervention. Serum markers, IL-6, Il-8, TNF-?, MCP-1, hs-CRP, leptin, TGFbeta, IL-1beta, and CRP will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Carpenter, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States